CLINICAL TRIAL: NCT03520283
Title: Use of Systems Support Mapping to Guide Patient-Driven Self-Management in Rural and Urban Cancer Survivors
Brief Title: Systems Support Mapping in Guiding Self-Management in Stage I-III Colorectal Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00048866; NCI-2018-00587 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 99118 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2018-04-12; First posted 2018-05-09 (Actual); Results first posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Cancer Survivor; Stage I Colorectal Cancer AJCC v8; Stage II Colorectal Cancer AJCC v8; Stage IIA Colorectal Cancer AJCC v8; Stage IIB Colorectal Cancer AJCC v8; Stage IIC Colorectal Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (MAP) (Experimental): Participants complete MAP in-clinic over 60-90 minutes.
  Interventions: Other: Interview; Other: Questionnaire Administration; Behavioral: System Support Mapping

INTERVENTIONS:
Other: Interview — Ancillary studies
Other: Questionnaire Administration — Ancillary studies
Behavioral: System Support Mapping — Complete MAP
  Other Names: MAP Intervention; System Support Mapping Intervention; MAP

SUMMARY:
This pilot trial studies how well systems support mapping works in guiding self-management in stage I-III colorectal cancer survivors. Systems support mapping helps participants to see complex self-management activities on paper, which makes them more actionable. Behavioral interventions, such as systems support mapping, may help colorectal cancer survivors facilitate self-awareness, create motivation for behavior change, and guide self-management.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the feasibility of the systems support mapping (MAP) intervention in colorectal cancer survivors, as characterized by enrollment, intervention adherence, and retention rates.

SECONDARY OBJECTIVES:

I. To evaluate intervention acceptability as characterized by participant ratings.

II. To describe outcome variability to inform future studies. III. To identify multi-level contextual factors influencing self-management (SM).

IV. To qualitatively assess feasibility, acceptability using semi-structured interviews.

V. To examine how study results vary by rural-urban context.

OUTLINE:

Participants complete MAP in-clinic over 60-90 minutes.

After completion of study, participants are followed-up for up to 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stage I-III colorectal cancer
* Within 2 years of completing active treatment for colorectal cancer
* Cognitively able to complete interviews as judged by the study team
* Able to understand, read and write English

Exclusion Criteria:

* Declined participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Sohl, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Derived] Sohl SJ, Befus D, Tooze JA, Levine B, Golden SL, Puccinelli-Ortega N, Pasche BC, Weaver KE, Lich KH. Feasibility of Systems Support Mapping to guide patient-driven health self-management in colorectal cancer survivors. Psychol Health. 2023 May;38(5):602-622. doi: 10.1080/08870446.2021.1979549. Epub 2021 Sep 27. PMID 34570677

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 66 people were approached to participate in this study. Only 24 were enrolled, 42 declined participation.
Groups:
- Enrolled Participants: Baseline characteristics of study participants that actually participated in study interventions.
- Declined Participants: Baseline characteristics of potential participants that declined participation
Period: Overall Study
Arm/Group | Enrolled Participants | Declined Participants
Started | 24 | 42
Completed | 24 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enrolled Participants | Declined Participants | Total
Number analyzed (Participants) | 24 | 42 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.91 (15.70) | 66.9 (11.29) | 63.90 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 22 | 37
  Male | 9 | 20 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 42 | 64
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 20 | 37 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 24 | 42 | 66
Marital Status [Count of Participants; unit: Participants] — Data only reported for participants who answered questions Population: Information was not collected for DECLINED PARTICIPANTS
  Participants
    Married or Living with Partner: number analyzed (Participants) | 23 | 0 | 23
    Married or Living with Partner | 13 |  | 13
    Separated/Divorced: number analyzed (Participants) | 23 | 0 | 23
    Separated/Divorced | 2 |  | 2
    Widowed/Single: number analyzed (Participants) | 23 | 0 | 23
    Widowed/Single | 8 |  | 8
Education Level [Count of Participants; unit: Participants] — Data only reported for participants who answered questions Population: Data only reported for participants who answered questions
  Participants
    Less than high school/High school graduate: number analyzed (Participants) | 23 | 0 | 23
    Less than high school/High school graduate | 3 |  | 3
    Technical school/Some college: number analyzed (Participants) | 23 | 0 | 23
    Technical school/Some college | 9 |  | 9
    College graduate/Post graduate degree: number analyzed (Participants) | 23 | 0 | 23
    College graduate/Post graduate degree | 11 |  | 11
Difficulty Paying Monthly Bills [Count of Participants; unit: Participants] — Data only reported for participants who answered questions Population: Data only reported for participants who answered questions
  Participants
    Very/somewhat difficult: number analyzed (Participants) | 22 | 0 | 22
    Very/somewhat difficult | 6 |  | 6
    Not very difficult: number analyzed (Participants) | 22 | 0 | 22
    Not very difficult | 11 |  | 11
    Not at all diffcult: number analyzed (Participants) | 22 | 0 | 22
    Not at all diffcult | 5 |  | 5
Confident in Filling Out Medical Forms (Health Literacy) [Count of Participants; unit: Participants] — Data only reported for participants who answered questions Population: Data only reported for participants who answered questions
  Participants
    Extremely/Quite a Bit: number analyzed (Participants) | 23 | 0 | 23
    Extremely/Quite a Bit | 20 |  | 20
    Somewhat/A Little Bit/Not at all: number analyzed (Participants) | 23 | 0 | 23
    Somewhat/A Little Bit/Not at all | 3 |  | 3
Times Received Income from AFDC, TANF, Work First, WIC or food stamps [Count of Participants; unit: Participants] — Data only reported for participants who answered questions Population: Data only reported for participants who answered questions
  Participants
    Never: number analyzed (Participants) | 23 | 0 | 23
    Never | 19 |  | 19
    Four times or less: number analyzed (Participants) | 23 | 0 | 23
    Four times or less | 3 |  | 3
    More than four times: number analyzed (Participants) | 23 | 0 | 23
    More than four times | 1 |  | 1
Rural Residence as Defined by Federal Office of Rural Health Policy (FORHP) [Count of Participants; unit: Participants] — Population: Information was not collected for DECLINED PARTICIPANTS.
  The FORHP accepts all non-Metro counties as rural and uses an additional method of determining rurality called the Rural-Urban Commuting Area (RUCA) codes. Like the MSAs, these are based on Census data that is used to assign a code to each Census Tract. Tracts inside Metropolitan counties with the codes 4-10 are considered rural.
  Participants
    Rural Residence as defined by FORHP: number analyzed (Participants) | 24 | 0 | 24
    Rural Residence as defined by FORHP | 5 |  | 5
    Not living in a rural residence: number analyzed (Participants) | 24 | 0 | 24
    Not living in a rural residence | 19 |  | 19
Use of Internet or Email [Count of Participants; unit: Participants] — Population: Information was no collected for DECLINED PARTICIPANTS.
  Participants
    Yes: number analyzed (Participants) | 24 | 0 | 24
    Yes | 22 |  | 22
    No: number analyzed (Participants) | 24 | 0 | 24
    No | 2 |  | 2
Cancer Type [Count of Participants; unit: Participants] — Population: Information was not collected for DECLINED PARTICIPANTS
  Participants
    Colon cancer: number analyzed (Participants) | 24 | 0 | 24
    Colon cancer | 17 |  | 17
    Rectal cancer: number analyzed (Participants) | 24 | 0 | 24
    Rectal cancer | 7 |  | 7
Summary Disease Stage at Diagnosis [Count of Participants; unit: Participants] — Part of the eligibility criteria were participants had to have a diagnosis of Stage I-III colorectal cancer based on the American Joint Committee on Cancer (AJCC) Tumor, lymph Nodes and Metastasis (TNM) system. The lower the stage number, the less the cancer has spread. Population: Information was not collected for DECLINED PARTICIPANTS
  Participants
    Stage I: number analyzed (Participants) | 24 | 0 | 24
    Stage I | 5 |  | 5
    Stage II: number analyzed (Participants) | 24 | 0 | 24
    Stage II | 7 |  | 7
    Stage III: number analyzed (Participants) | 24 | 0 | 24
    Stage III | 12 |  | 12
Recurrent Disease [Count of Participants; unit: Participants] — Population: Information was not collected for DECLINED PARTICIPANTS
  Participants
    Yes: number analyzed (Participants) | 24 | 0 | 24
    Yes | 0 |  | 0
    No: number analyzed (Participants) | 24 | 0 | 24
    No | 24 |  | 24
Underwent Surgery [Count of Participants; unit: Participants] — Population: Information was not collected for DECLINED PARTICIPANTS
  Participants
    Yes: number analyzed (Participants) | 24 | 0 | 24
    Yes | 23 |  | 23
    No: number analyzed (Participants) | 24 | 0 | 24
    No | 1 |  | 1
Received Radiation [Count of Participants; unit: Participants] — Population: Information was not collected for DECLINED PARTICIPANTS
  Participants
    Yes: number analyzed (Participants) | 24 | 0 | 24
    Yes | 9 |  | 9
    No: number analyzed (Participants) | 24 | 0 | 24
    No | 15 |  | 15
Received Chemotherapy [Count of Participants; unit: Participants] — Population: Information was not collected for DECLINED PARTICIPANTS
  Participants
    Yes: number analyzed (Participants) | 24 | 0 | 24
    Yes | 17 |  | 17
    No: number analyzed (Participants) | 24 | 0 | 24
    No | 7 |  | 7
Number of Comorbidities (Range 0-14) [Median (Full Range); unit: median of comorbidities of participants] — Population: Information was not collected for DECLINED PARTICIPANTS
  median of comorbidities of participants
    number analyzed (Participants) | 24 | 0 | 24
    (all) | 1 [0 to 5] |  | 1 [0 to 5]
Months Since Last Cancer Treatment [Median (Full Range); unit: months] — Population: Information was not collected for DECLINED PARTICIPANTS
  months
    number analyzed (Participants) | 24 | 0 | 24
    (all) | 9 [1 to 21] |  | 9 [1 to 21]
Minutes Traveled to Clinic [Median (Full Range); unit: minutes] — Population: Information was not collected for DECLINED PARTICIPANTS
  minutes
    number analyzed (Participants) | 24 | 0 | 24
    (all) | 34 [10 to 150] |  | 34 [10 to 150]

OUTCOME MEASURES:

1. Primary Outcome: Enrollment Rate
Description: To be calculated as the percent of eligible participants approached who agree to participate. Will use one-sample tests of negative binomial probabilities and binomial proportions to compare rates of feasibility to hypothesized values. Rates will be summarized using point estimates and 95% confidence intervals.
Time Frame: Up to 1 year
Population: Out of 66 participants asked to participate, only 24 were eligible/enrolled into the intervention.
Measure: Number (95% Confidence Interval); unit: Percent probability of participants
Groups:
- Enrollment Rate - Eligible Participants: To be calculated as the percent of eligible participants approached who agree to participate. Will use one-sample tests of negative binomial probabilities and binomial proportions to compare rates of feasibility to hypothesized values. Rates will be summarized using point estimates and 95% confidence intervals.
Arm/Group | Enrollment Rate - Eligible Participants
Number analyzed (Participants) | 66
Percent probability of participants | 0.36 [0.25 to 0.49]

2. Primary Outcome: Participation Rate
Description: To be calculated as the percent of participants who complete the study intervention among those enrolled. Will use one-sample tests of negative binomial probabilities and binomial proportions to compare rates of feasibility to hypothesized values. Rates will be summarized using point estimates and 95% confidence intervals.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Measure: Number (95% Confidence Interval); unit: percentage of completed intervention
Groups:
- Participation Rate - Eligible Participants: To be calculated as the percent of participants who complete the study intervention among those enrolled. Will use one-sample tests of negative binomial probabilities and binomial proportions to compare rates of feasibility to hypothesized values. Rates will be summarized using point estimates and 95% confidence intervals.
Arm/Group | Participation Rate - Eligible Participants
Number analyzed (Participants) | 24
percentage of completed intervention | 0.88 [0.68 to 0.97]

3. Primary Outcome: Retention Rate
Description: To be calculated as the proportion of participants who complete the study measures among those enrolled. Will use one-sample tests of negative binomial probabilities and binomial proportions to compare rates of feasibility to hypothesized values. Rates will be summarized using point estimates and 95% confidence intervals.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Measure: Mean (95% Confidence Interval); unit: proportion of completed study measures
Groups:
- Retention Rate - Eligible Participants: To be calculated as the number of participants who complete the study measures among those enrolled. Will use one-sample tests of negative binomial probabilities and binomial proportions to compare rates of feasibility to hypothesized values. Rates will be summarized using point estimates and 95% confidence intervals.
Arm/Group | Retention Rate - Eligible Participants
Number analyzed (Participants) | 24
proportion of completed study measures | 0.83 [0.63 to 0.95]

4. Secondary Outcome: Self-reported Ratings of Intervention Acceptability
Description: Descriptive statistics will be used to summarize participant ratings of acceptability of intervention.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Population: 20 out of 24 participants were assessed at follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Self-reported Ratings of Intervention Acceptability - Eligible Participants: Descriptive statistics will be used to summarize participant ratings of acceptability.
Arm/Group | Self-reported Ratings of Intervention Acceptability - Eligible Participants
Number analyzed (Participants) | 20
Participants
  Liked the intervention quite a bit/very much | 16
  Liked the intervention a little bit/somewhat | 4
  Found intervention helpful very much/quite a bit | 15
  Found intervention helpful a little bit/somewhat | 5
  Would continue to use what they learned quite a bit/very much | 18
  Would continue to use what they learned a little bit/somewhat | 2
  Found interventionist competent and sensitive quite a bit/very much | 20

5. Secondary Outcome: Measures of Autonomy Assessed by Index of Autonomous Functioning
Description: Each item in the scale ranges from 0-5, where 0=not at all true and 5=completely true. Scale is a mean of these items and thus ranges from the same minimum of 0 to the same maximum of 5. A higher score represent higher degree of autonomy.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Measures of Autonomy Assessed by Index of Autonomous Functioning: Autonomy will be assessed at baseline and at 2 weeks with a difference of the two time points.
Arm/Group | Measures of Autonomy Assessed by Index of Autonomous Functioning
Number analyzed (Participants) | 24
score on a scale
  Baseline | 4.4 (0.6)
  Two weeks | 4.7 (0.4)
  Difference in time points | 0.4 (0.6)

6. Secondary Outcome: Self-efficacy for Managing Cancer - Chronic Disease Scale
Description: Scale is a mean of physical and emotional functional management of chronic disease. Each of which runs from 1 (not at all confident) to 10 (totally confident). A higher score represents a higher degree of confidence in self-efficacy.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Self-efficacy for Managing Cancer - Chronic Disease Scale: Self-efficacy for managing cancer will be assessed as a mean value at baseline and at two weeks with a difference of values between the two time points.
Arm/Group | Self-efficacy for Managing Cancer - Chronic Disease Scale
Number analyzed (Participants) | 24
score on a scale
  Baseline | 7.7 (2.1)
  Two weeeks | 8.6 (1.5)
  Difference between the two time points | 0.6 (1.2)

7. Secondary Outcome: Self-Efficacy for Managing Symptoms - Patient Reported Outcomes Measurement Information System (PROMIS) Short Form
Description: Overall score is based emotional and physical management of symptoms and is converted to a norm-based score that ranges from 0-100. Higher score means more of construct or response of managing symptoms.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Self-Efficacy for Managing Symptoms - (PROMIS) Short Form: Self-efficacy for managing cancer will be assessed as a mean value at baseline and at two weeks with a difference of values between the two time points.
Arm/Group | Self-Efficacy for Managing Symptoms - (PROMIS) Short Form
Number analyzed (Participants) | 24
score on a scale
  Baseline | 49.8 (8.4)
  Two weeeks | 55.2 (8.6)
  Difference between the two time points | 4.3 (7.4)

8. Secondary Outcome: PROMIS - Relatedness Assessed by Healing Encounters and Attitudes Lists (HEAL) Patient-Provider Connection
Description: The overall score is based on participant's relatedness to interventionists and is converted to a norm-based score that ranges from 26.6-72.5. Higher score on the HEAL measure means a higher degree of patient-provider connection as assessed by the patient.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- PROMIS - Relatedness Assessed by Healing Encounters and Attitudes Lists Patient-Provider Connection: Relatedness to interventionists was measured at 2 weeks after intervention.
Arm/Group | PROMIS - Relatedness Assessed by Healing Encounters and Attitudes Lists Patient-Provider Connection
Number analyzed (Participants) | 24
score on a scale | 66.2 (7.5)

9. Secondary Outcome: Psychological Stress Assessed by Perceived Stress Scale
Description: Descriptive statistics (means, standard deviations) will be used to summarize proximal outcomes and change in health outcomes by assessment measure. The primary interest will be in estimating the variance for use in planning future studies. A 4-item questionnaires to assess participants' stress during the intervention at baseline and at two weeks with a difference of both time points. Scoring scale is from 0-4 ( 0 - never and 4 - very often). Scoring range is 0-16 with the higher score indicating higher stress.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Psychological Stress Assessed by Perceived Stress Scale - Eligible Participants: Descriptive statistics (means, standard deviations) will be used to summarize proximal outcomes and change in health outcomes by assessment measure. The primary interest will be in estimating the variance for use in planning future studies.
Arm/Group | Psychological Stress Assessed by Perceived Stress Scale - Eligible Participants
Number analyzed (Participants) | 24
score on a scale
  Baseline | 8.1 (1.9)
  Two weeks | 6.7 (2.9)
  Difference in both time points | -1.0 (2.2)

10. Secondary Outcome: Symptoms Assessed by Patient-Reported Outcomes Measurement Information System (PROMIS) Profile 29
Description: PROMIS instruments contain a fixed number of items from seven PROMIS domains: depression; anxiety; physical function; pain interference; fatigue; sleep disturbance; and ability to participate in social roles and activities. The PROMIS-29, a generic health-related quality of life survey, assesses each of the 7 PROMIS domains with 4 questions. The questions are ranked on a 5-point Likert Scale. There is also one 11-point rating scale for pain intensity. Norm-based scores have been calculated for each domain on the PROMIS measures, so that a score of 50 represents the mean or average of the reference population. A score of 60 means that the person is one standard deviation above the reference population. On symptom oriented domains of PROMIS-29 (anxiety, depression, fatigue, pain interference, and sleep disturbance), higher scores represent worse symptomatology. On the function oriented domains (physical functioning and social role) higher scores represent better functioning.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Population: Not all eligible participants may have completed the intervention. The difference scores are computed only on the n=20 (or 18) who have *both* scores, which is why the difference scores are different from simply taking the difference of the 2 reported means
Measure: Mean (Standard Deviation); unit: T-score on a scale
Groups:
- Symptoms Assessed by PROMIS Profile 29 - Eligible Participants: Descriptive statistics (means, standard deviations) will be used to summarize proximal outcomes and change in health outcomes by assessment measure. The primary interest will be in estimating the variance for use in planning future studies.
Arm/Group | Symptoms Assessed by PROMIS Profile 29 - Eligible Participants
Number analyzed (Participants) | 24
T-score on a scale
  Physical Function - Baseline | 46.0 (8.5)
  Physical Function at Follow-Up: number analyzed (Participants) | 20
  Physical Function at Follow-Up | 47.3 (10.4)
  Physical Function - Difference between the two time points: number analyzed (Participants) | 20
  Physical Function - Difference between the two time points | 0.2 (6.5)
  Anxiety - Baseline: number analyzed (Participants) | 23
  Anxiety - Baseline | 50.3 (8.8)
  Anxiety at Follow-Up: number analyzed (Participants) | 20
  Anxiety at Follow-Up | 46.4 (8.5)
  Anxiety - Difference between the two time points: number analyzed (Participants) | 20
  Anxiety - Difference between the two time points | -2.3 (6.7)
  Depression - Baseline | 47.1 (7.7)
  Depression at Follow-Up: number analyzed (Participants) | 20
  Depression at Follow-Up | 45.3 (6.1)
  Depression - Difference between the two time points: number analyzed (Participants) | 20
  Depression - Difference between the two time points | -0.1 (5.7)
  Fatigue - Baseline | 51.9 (10.15)
  Fatigue at Follow-Up: number analyzed (Participants) | 20
  Fatigue at Follow-Up | 46.2 (9.4)
  Fatigue - Difference between the two time points: number analyzed (Participants) | 20
  Fatigue - Difference between the two time points | -4.7 (6.9)
  Sleep Disturbance - Baseline | 52.1 (7.8)
  Sleep Disturbance at Follow-Up: number analyzed (Participants) | 20
  Sleep Disturbance at Follow-Up | 49.3 (9.3)
  Sleep Disturbance - Difference between the two time points: number analyzed (Participants) | 20
  Sleep Disturbance - Difference between the two time points | -1.8 (6.3)
  Social Roles - Baseline | 50.1 (8.3)
  Social Roles at Follow-Up: number analyzed (Participants) | 18
  Social Roles at Follow-Up | 52.0 (10.6)
  Social Roles - Difference between the two time points: number analyzed (Participants) | 18
  Social Roles - Difference between the two time points | 1.6 (8.9)
  Pain Interference - Baseline | 52.4 (9.5)
  Pain Interference at Follow-Up: number analyzed (Participants) | 20
  Pain Interference at Follow-Up | 51.4 (10.0)
  Pain Interference - Difference between the two time points: number analyzed (Participants) | 20
  Pain Interference - Difference between the two time points | -0.9 (7.2)
  Pain Intensity - Baseline | 3.0 (2.8)
  Pain Intensity at Follow-Up: number analyzed (Participants) | 20
  Pain Intensity at Follow-Up | 2.5 (2.6)
  Pain Intensity - Difference between the two time points: number analyzed (Participants) | 20
  Pain Intensity - Difference between the two time points | -0.6 (1.7)

11. Secondary Outcome: Health Behaviors Assessed by Items on Tobacco Use
Description: Descriptive statistics will be used to summarize proximal outcomes. Participants were asked questions about their health behavior related to their past or present smoking behaviors (i.e. packs per day, last time they smoked) in order to help improve upon the information received to offer support for future studies.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Measure: Count of Participants; unit: Participants
Groups:
- Health Behaviors - Tobacco Use: Participants' status of tobacco use will be assessed during at baseline survey.
Arm/Group | Health Behaviors - Tobacco Use
Number analyzed (Participants) | 24
Participants
  Ever-smokers | 6
  Never smokers | 18
  Last cigarette more than 1 year ago prior to baseline survey | 6

12. Secondary Outcome: Qualitative Assessment of Feasibility With Semi-structured Interviews
Description: Will conduct a qualitative content analysis. Qualitative data will be sent to an external vendor to be transcribed. Two internal study team members will double-code at least 10% of coding of transcripts from the semi-structured interviews and resolve any disagreements to ensure that robust and unbiased results are achieved. Will evaluate qualitative and quantitative analyses in a mixed-methods framework for consistency and discrepancies across all analyses to refine the protocol.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Population: Qualitative interview data was collected from 19 participants. Information gained related to study processes enhanced understanding of quantitative results and will inform the next phase of study
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 24
Participants | 19

13. Secondary Outcome: Qualitative Analysis of Systems Support Maps
Description: The internal study team will work with collaborators through an iterative process to facilitate a qualitative content analysis of the large quantity of textual MAP data. Will examine all qualitative analyses by urban-rural status as classified using Rural Urban Commuting Area Codes. Qualitative results will be summarized by urban-rural status. Will also compare MAP results by rural-urban status.
Time Frame: Up to 1 year
Population: Textual data from the intervention mapping was collected from 21 participants. Content analysis identified multi-level contextual factors influencing self-management and results were examined by rural-urban status.
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 24
Participants | 21

14. Secondary Outcome: Health Behaviors Assessed by Items on Physical Activity
Description: Participant's ability to participate in physical activities (types of activities, intensity, etc.) will be assessed. Descriptive statistics will be used to summarize proximal outcomes. The primary interest will be in estimating the variance for use in planning future studies.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Population: Not all participants may have completed the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 24
Participants
  Rarely or never do any physical activity - Baseline: number analyzed (Participants) | 23
  Rarely or never do any physical activity - Baseline | 3
  Rarely or never do any physical activity - At two weeks: number analyzed (Participants) | 19
  Rarely or never do any physical activity - At two weeks | 3
  Do some light/moderate physical activity but not every week - Baseline | 7
  Do some light/moderate physical activity but not every week - At two weeks: number analyzed (Participants) | 19
  Do some light/moderate physical activity but not every week - At two weeks | 4
  Light physical activity every week - Baseline: number analyzed (Participants) | 23
  Light physical activity every week - Baseline | 16
  Light physical activity every week - At two weeks: number analyzed (Participants) | 20
  Light physical activity every week - At two weeks | 15
  Moderate physical activity every week but less than 30 minutes a day or 5 days a week - Baseline: number analyzed (Participants) | 23
  Moderate physical activity every week but less than 30 minutes a day or 5 days a week - Baseline | 11
  Moderate physical activity every week but less than 30 minutes a day or 5 days a week - At two weeks: number analyzed (Participants) | 19
  Moderate physical activity every week but less than 30 minutes a day or 5 days a week - At two weeks | 10
  Vigorous activity every week but less than 20 minutes a day or three days a week - Baseline: number analyzed (Participants) | 23
  Vigorous activity every week but less than 20 minutes a day or three days a week - Baseline | 4
  Vigorous activity every week but less than 20 minutes a day or three days a week - At two weeks: number analyzed (Participants) | 19
  Vigorous activity every week but less than 20 minutes a day or three days a week - At two weeks | 2
  30 minutes or more of moderate activity five or more days a week - Baseline: number analyzed (Participants) | 23
  30 minutes or more of moderate activity five or more days a week - Baseline | 6
  30 minutes or more of moderate activity five or more days a week - At two weeks: number analyzed (Participants) | 19
  30 minutes or more of moderate activity five or more days a week - At two weeks | 8
  20 min or more of vigorous activity 3 or more days a week - Baseline: number analyzed (Participants) | 23
  20 min or more of vigorous activity 3 or more days a week - Baseline | 4
  20 min or more of vigorous activity 3 or more days a week - At two weeks: number analyzed (Participants) | 19
  20 min or more of vigorous activity 3 or more days a week - At two weeks | 2

15. Secondary Outcome: Health Behaviors Assessed by Items on Use of Complementary Health Approaches
Description: Participants will assess the use of complementary or alternative therapies use since first diagnosed with cancer. Descriptive statistics will be used to summarize proximal outcomes. The primary interest will be in estimating the variance for use in planning future studies.
Time Frame: Approximately 1.5-2 hours at baseline visit in clinic with a 2-week follow-up 2 weeks later
Population: Not all participants completed interventions in the two week (follow up) time frame
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 24
Participants
  Special Diets in the past year | 3
  Special Diets in the past two weeks: number analyzed (Participants) | 20
  Special Diets in the past two weeks | 3
  Natural Products in the past year | 4
  Natural products in the past two weeks: number analyzed (Participants) | 20
  Natural products in the past two weeks | 4
  Mind/body therapies in the past year | 8
  Mind/body therapies in the past two weeks: number analyzed (Participants) | 20
  Mind/body therapies in the past two weeks | 5
  Personal prayer in past year | 14
  Personal prayer in the past two weeks: number analyzed (Participants) | 20
  Personal prayer in the past two weeks | 12
  Other stress support in the past year | 1
  Other stress support in the past two weeks: number analyzed (Participants) | 20
  Other stress support in the past two weeks | 2

16. Secondary Outcome: Qualitative Assessment of Acceptability With Semi-structured Interviews
Description: as for outcome 12
Time Frame: Up to 1 year
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 24
Participants | 19

17. Secondary Outcome: Qualitative Assessment of Changes in Outcomes With Semi-structured Interviews
Description: as for outcome 12
Time Frame: Up to 1 year
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Enrolled Participants
Number analyzed (Participants) | 24
Participants | 19

ADVERSE EVENTS:
Time Frame: Two weeks following the intervention
Arm/Group | Supportive Care (MAP)
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 2/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (MAP) (N=24)
Tearfulness (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-07): https://cdn.clinicaltrials.gov/large-docs/83/NCT03520283/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT03520283/ICF_001.pdf